CLINICAL TRIAL: NCT05638581
Title: Trauma Resuscitation With Low-Titer Group O Whole Blood or Products
Acronym: TROOP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jan O. Jansen, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1UG3HL157401-01A1 (NIH); 1UG3HL157401-01A1 (NIH); 1U24HL157310-01A1 (NIH)
Record Dates: First submitted 2022-11-08; First posted 2022-12-06 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Wounds and Injuries; Shock, Hemorrhagic
Keywords: Massive Transfusion; Trauma; Shock; Hemorrhage; Plasma; Platelets; Red Blood Cells; Low-Titer Group O Whole Blood; Blood components
MeSH Terms: conditions — Wounds and Injuries; Shock, Hemorrhagic; Shock; Hemorrhage | interventions — Elements

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Care providers will be blinded to assignment until the point of randomization, which is when the cooler is opened, in the trauma bay, to remove blood products for transfusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LTOWB (Active Comparator): Participants randomized to receive (Low Titer O Whole Blood [LTOWB])
  Interventions: Biological: LTOWB
- Components (Active Comparator): Participants randomized to receive the component blood products.
  Interventions: Biological: Components

INTERVENTIONS:
Biological: LTOWB — Participants will receive Low Titer O Whole Blood administered intravenously or intraosseously.
  Arms: LTOWB
Biological: Components — Participants will receive separated blood components (i.e., units of red cells, plasma, platelets, and cryoprecipitate) co-administered intravenously or intraosseously.
  Arms: Components

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of unseparated whole blood (referred to as Low-Titer Group O Whole Blood) and the separate components of whole blood (including red cells, plasma, platelets, and cryoprecipitate) in critically injured patients who require large-volume blood transfusions.

DETAILED DESCRIPTION:
Trauma is one of the leading causes of death in the United States, and disproportionately affects the young, killing those who might otherwise have lived long and productive lives. Injuries account for more years of potential life lost before age 75 than any other cause. Hemorrhage remains the most common cause of preventable death after injury, and blood transfusion is an essential part of treatment. Modern blood banking practices separate donated whole blood into components. The current standard of care in trauma transfusion is the balanced administration of equal numbers of units of blood components (packed red blood cells, plasma, and platelets), effectively attempting to reconstitute whole blood. A renewed approach to blood transfusion therapy in trauma is to use whole blood from the outset, which has not been separated. Compared with component therapy, whole blood offers several potential advantages, but there are only a small number of, mostly observational, studies comparing whole blood and component therapy, and they are very heterogeneous.

The TROOP trial will include injured adults with hemorrhagic shock anticipated to require massive blood transfusions, who will be randomized to receive either whole blood (LTOWB) or blood components. This will allow a direct comparison to see if one type of transfusion is more strongly associated with improved clinical outcomes over the other.

The knowledge gained from this clinical trial will transform the way in which massively bleeding trauma patients are transfused. The trial is exceedingly well positioned to improve mortality from trauma and reduce the number of preventable deaths resulting from hemorrhagic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Adult trauma patient (estimated age > 15 or weight > 50 kg, if age unknown)
2. Patient taken to trauma center directly from scene
3. Commencement of blood transfusion (PRBC, plasma or LTOWB), in pre-hospital or in-hospital setting
4. Activation of site-specific Massive Hemorrhage Protocol or Massive Transfusion Protocol
5. Traumatic injury with at least one of the following:

   1. Confirmed or suspected acute major bleeding
   2. Assessment of Blood Consumption (ABC) Score ≥2

Exclusion Criteria:

1. Patients who have received, prehospital or in-hospital more than two units of LTOWB; the equivalent in components (two units of packed red blood cells and two units of plasma); or a combination of the two (more than one unit of LTOWB, one unit of packed cells, and one unit of plasma). Most trauma centers hold two units of either packed red blood cells (with two units of plasma) or two units of LTOWB in the emergency department. This stock is used to initiate transfusion, while the massive hemorrhage protocol is activated from the blood bank.
2. Patients transferred from another hospital
3. Children <15 years (in most communities, patients aged 15-18 years are treated at adult trauma centers, and patients in this age group frequently suffer life-threatening injuries, and will therefore be included)
4. Known prisoners, defined as individuals involuntarily confined or detained in a penal institution (including juvenile detention, involuntary psychiatric commitment, or court-ordered residential substance abuse treatment)
5. Moribund patients expected to die within 1 hour
6. Patients who required an ED thoracotomy or received more than 5 consecutive minutes of cardiopulmonary resuscitation (prior to receiving randomized blood products)
7. Patients with known "do not resuscitate" orders prior to randomization
8. Patients who refuse the administration of blood products
9. Individuals with a research "opt out" bracelet.
10. Greater than 20% total body surface area (TBSA) burns
11. Suspected inhalation injury victims
12. Patients who are obviously pregnant on clinical examination or known to be pregnant as provided by the subject or legally authorized representative

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
6-hour Mortality | First 6 hours after randomization
  Participant vital status at 6-hours following randomization (randomization defined as product container is opened for administration to participant)

SECONDARY OUTCOMES:
24-hour Mortality | First 24 hours after randomization
  Participant vital status at 24-hours following randomization
Hospital/30-day Mortality | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  Participant vital status at hospital discharge or 30-days post randomization (whichever the earlier)
Incidence of Pre-specified Complications | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  The number of participants experiencing pre-specified complications. Pre-specified complications include: Acute kidney injury; Ventilator-associated pneumonia; Multiorgan failure; Transfusion-related hyperkalemia; Transfusion-related hypocalcemia; Transfusion associated circulatory overload; Acute respiratory distress syndrome; Symptomatic and asymptomatic deep vein thrombosis; Symptomatic and asymptomatic pulmonary embolism; Bleeding after hemostasis requiring intervention; Stroke; Myocardial infarction; Abdominal compartment syndrome; Transfusion-related allergic reactions; Febrile non-hemolytic transfusion reaction; Systemic inflammatory response syndrome; Sepsis; Alloimmunization in women of childbearing age
Adjudicated Primary Cause of Death | 30-days post randomization
  Primary cause of death as reviewed and determined by the study investigators (consensus)
Length of Stay (Hospital and Intensive Care Unit) | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  Number of hours hospitalized (includes both hospital and intensive care unit time)
Hospital-, Ventilator- and Intensive Care Unit-free days | 30-days post randomization
  Number of days participant was alive and out of the hospital; number of days participant was not on a ventilator; and the number of days the participant was not in the intensive care unit.
Incidence of major surgical procedures | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  The proportion of participants undergoing major surgical procedures.
Time to hemostasis in those undergoing procedures with a hemostatic component | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  Time to hemostasis refers to the time that the subject achieved hemorrhage control (anatomic hemostasis and resuscitation complete) following emergency department arrival.
Number and type of blood products used until hemostasis is achieved and from hemostasis to 24 hours after randomization | First 24 hours after randomization
  The number of units and type of blood products (e.g. whole blood, packed red blood cells, platelets, plasma, etc.)
Discharge destination | At hospital discharge or 30-days post randomization (whichever the earlier)
  Discharge destination will be measured as a categorical variable. Categories will be tallied and compared between the two study arms. Example variables include: discharged to home, discharged to another primary care facility, discharged to hospice, etc.
Functional status | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  Functional status will be measured by Extended Glasgow Outcome Scale (GOSE). The GOSE is a tool used to measure recovery following brain injury and assists with prediction of long-term rehabilitation. The 8 scoring categories are death, vegetative state, lower severe disability, upper severe disability, lower moderate disability, upper moderate disability, lower good recovery and upper good recovery. A higher GOSE score correlates with better outcome.
Patient's quality of life | From randomization to hospital discharge or 30-days post randomization (whichever the earlier)
  Quality of life will be measured by the Euroqol Group's EQ-5D quality of life measurement. The EQ-5D is a patient-reported questionnaire assessing health status in terms of five dimensions of health (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression). Lower EQ-5D scores are associated with better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jansen, MBBS, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, UAB Hospital, Birmingham, Alabama
  - Los Angeles County + University of Southern California (LAC + USC) Medical Center, Los Angeles, California
  - University Medical Center New Orleans LCMC Health, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oregon Health and Sciences University Hospital, Portland, Oregon
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center Houston, Houston, Texas
  - University of Texas Health San Antonio and University Health System, San Antonio, Texas
  - Harborview Medical Center, Seattle, Washington
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansen JO, Pedroza C, Novelo LL, Hao T, DeWildt GR, Coton CF, Mansoor K, Stephens SW, Marques MB, Stubbs JR, Richter JR, Wang HE, Holcomb JB, DeSantis SM. Trauma resuscitation with Low-Titer Group O Whole Blood Or Products: study protocol for a randomized clinical trial (the TROOP trial). Trials. 2025 Aug 2;26(1):266. doi: 10.1186/s13063-025-08971-y. PMID 40753420
- [Derived] Meizoso JP, Cotton BA, Lawless RA, Kodadek LM, Lynde JM, Russell N, Gaspich J, Maung A, Anderson C, Reynolds JM, Haines KL, Kasotakis G, Freeman JJ. Whole blood resuscitation for injured patients requiring transfusion: A systematic review, meta-analysis, and practice management guideline from the Eastern Association for the Surgery of Trauma. J Trauma Acute Care Surg. 2024 Sep 1;97(3):460-470. doi: 10.1097/TA.0000000000004327. Epub 2024 Mar 27. PMID 38531812
- See also: TROOP Consortium website — http://trooptrial.org